CLINICAL TRIAL: NCT05040932
Title: A First-In-Human, Multicenter, Open-Label, Phase I Dose Escalation Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of YH004 As A Single Agent And Combination With Toripalimab In Subjects With Advanced Solid Tumors And Relapsed Or Refractory Non-Hodgkin Lymphoma
Brief Title: Study of YH004 (4-1BB Agonist Antibody) in Advanced or Metastatic Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH004002
Record Dates: First submitted 2021-08-27; First posted 2021-09-10 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Eucure; YH004; anti-4-1BB; Toripalimab; anti-PD-1
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YH004 (Experimental): The dose escalation phase includes 7 dose levels of YH004, and the highest dose is up to 10mg/kg. Route of administration is IV infusion, and the frequency of administration is once every 3 weeks (Q3W). one cycle is 3 weeks, and treatment can be up to 16 cycles if patients receive benefits.
  Interventions: Drug: YH004

INTERVENTIONS:
Drug: YH004 — IV infusion once every 3 weeks (Q3W).

SUMMARY:
YH004 is a humanized monoclonal antibody that specifically binds to 4-1BB, and acts as an agonist against 4-1BB.

This first in human study of YH004 is designed to establish the maximum tolerated dose (MTD) and/or the recommended Phase II dose (RP2D) of YH004, both as a single agent (monotherapy) and in combination with a fixed dose of anti-PD-1 antibody (Toripalimab) in the treatment of advanced solid tumors and relapsed or refractory non-Hodgkin Lymphoma.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, two-stage, FIH Phase 1 study, utilizing an accelerated dose escalation followed by a traditional 3 + 3 dose escalation algorithm to identify the MTD and/or RP2D of YH004 as a single agent (monotherapy) and in combination with Toripalimab. The first stage of the study is the dose escalation phase (i.e., Phase 1a). The second stage of the study is the dose expansion phase (i.e., Phase 1b). During the study, dose interruption(s) and/or delay(s) may be implemented based on toxicity. Dose modifications are permitted following protocol guidelines. Intra-patient dose escalations will be allowed for the early dose cohorts (single-patient dose groups) in Phase 1a. Patients will be considered evaluable for safety and tolerability if they receive at least one dose of YH004 or Toripalimab at the specified cohort dose. Patients in all parts of the trial will remain on therapy until confirmed disease progression or for 1 year, whichever occurs first. However, patients who are clinically unstable will discontinue following the initial assessment of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years to 80 years at the time of screening.
* Ability to understand and willingness to sign a written informed consent document.
* Subjects must have advanced histologically or cytologically confirmed solid tumor or relapsed or refractory Non-Hodgkin lymphoma.
* Adequate bone marrow, liver, and renal functions.
* Men and women of childbearing potential must agree to take highly effective contraceptive methods.
* Women of reproductive potential must have negative serum beta human chorionic gonadotropin (β -HCG) pregnancy test within 7 days of the first dose.

Exclusion Criteria:

* Receipt of systemic anticancer therapy including investigational agents or devices within 5 half-lives of the first dose of study treatment.
* Known active CNS metastasis.
* Has received a live-virus vaccine within 28 days.
* History of clinically significant sensitivity or allergy to monoclonal antibodies and their excipients or known allergies to antibodies produced from Chinese hamster ovary cells.
* Abnormality of QT interval or syndrome.
* Patients with history of Grade ≥ 3 immune-related AEs (irAEs) or irAE.
* Patients who receive concurrent or prior use of an immunosuppressive agent within 4 weeks of the first dose of study drug.
* Previous exposure to anti-CD137 (eg, utomilumab, urelumab) antibodies. .
* Active or chronic autoimmune disease that has required systemic treatment in the past 3 years or who are receiving systemic therapy for an autoimmune or inflammatory disease.
* Has a clinically significant cardiac condition, including unstable angina, acute myocardial infarction within 6 months.
* Has an active infection before the first dose of study treatment.
* History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis, or history of interstitial lung disease..
* Female patients who are pregnant or breastfeeding.
* Any evidence of severe or uncontrolled systemic disease.
* Any condition that the investigator or primary physician believes may not be appropriate for participating the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2023-07-16 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) including determination of DLTs and serious AEs (SAEs) | up to 24 months
  Adverse events will be assessed, and severity will be assigned by using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Maximum tolerated dose (MTD) and/or the recommended Phase II dose (RP2D) | up to 24 months
  The MTD and/or RP2D will be determined based on TEAEs

CONTACTS AND LOCATIONS:
Overall Officials: Rong Chen, Ph.D, Study Chair — Eucure (Beijing) Biopharma Co., Ltd
Locations (3):
- Australia (3):
  - Cabrini Health Limited, Malvern East
  - Westmead Hospital, Sydney
  - Southside Cancer Care Centre, School of Medicine, University of Wollongong, Wollongong